CLINICAL TRIAL: NCT00974740
Title: DIATOR - Diabetes Intervention With Atorvastatin. A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Effect of Atorvastatin on Residual Beta-cell Function and Glycemic Control in Patients With Newly Diagnosed Type 1 Diabetes Mellitus
Brief Title: DIATOR-Diabetes Intervention With Atorvastatin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: for lack of recruitment
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33/0136-Diator
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- atorvastatin matching placebo (Placebo Comparator): atorvastatin matching placebo
  Interventions: Drug: atorvastatin matching placebo
- atorvastatin (Experimental): 40 mg atorvastatin for 4 weeks (run-in period), then 80 mg atorvastatin, total treatment period was 18 months
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 40 mg (tablet for oral intake) once daily in the evening for 4 weeks, thereafter 80 mg for the remaining treatment period (total treatment period 18 months)
  Other Names: Sortis
  Arms: atorvastatin
Drug: atorvastatin matching placebo — atorvastatin matching placebo tablets once daily in the evening, corresponding to 40 mg atorvastatin for the first 4 weeks (run-in period), and corresponding to 80 mg atorvastatin thereafter (total treatment period 18 months)
  Arms: atorvastatin matching placebo

SUMMARY:
Clinical studies have shown that immunomodulators (like Anti-CD3 antibodies) have effects on beta-cell-preservation. The lipid-lowering agent atorvastatin is also a potent immunomodulator. In this study the effects of 80 mg atorvastatin per day on preservation of beta-cell function in recent onset type 1 diabetes were studied, as determined by stimulated C-peptide levels.

DETAILED DESCRIPTION:
The objectives of this study were as follows:

* To assess the effect of atorvastatin on pancreatic beta-cell function as measured by C-peptide after a liquid mixed meal stimulation in patients with newly diagnosed type 1 diabetes,
* To assess the effect on metabolic control as measured by HbA1c and insulin requirements,
* To assess safety and tolerability of atorvastatin in subjects with newly diagnosed type 1 diabetes,
* To assess the effect on risk factors of diabetic complications as indicated by changes in lipids and CRP, and
* To assess the effect on systemic immune abnormalities as measured by effects on beta-cell autoantibodies, blood cytokines and chemokines on protein and transcriptional level.

Study duration: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Insulin treated patients with a newly diagnosed type 1 diabetes mellitus as defined by the ADA criteria at least two weeks but not later than 3 months after start of insulin treatment
* Age 18 to 39 years, inclusive
* Male patient or female patient using adequate contraceptive methods
* Tested positive for at least one of the three islet autoantibodies GAD65, IA2 or ICA

Exclusion Criteria:

* History of a malignancy
* Presence of a clinically significant hepatic or renal disease, as indicated, but not limited to a serum creatinine elevated more than ten percent above the upper limit of normal, elevation of AST or ALT more than 3 times the upper limit of normal
* Any other acute or chronic condition that may affect the patient's response to treatment or might be associated with an increased risk for the patient to participate, as judged by the investigator
* Current use of anti-inflammatory or immunomodulatory drugs, antihypertensive, lipid-lowering, or antidiabetic drugs other than insulin
* Pregnant or nursing women or women intending to become pregnant
* Known or suspected allergy to atorvastatin or any component of thr trial product
* Known myopathy, myalgia or myositis with a serum-CPK above 3 times the upper limit of normal
* Patients who had a severe blood loss (>= 400 mL, e.g. blood donation) within 2 months prior to visit 2
* Any significant laboratory abnormality
* A serum LDL-cholesterol above 150 mg/dL at time of screening
* Unwillingness to comply with study procedures

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
C-peptide after a liquid mixed meal stimulation | at randomization, after 12 months, and after 18 months of treatment

SECONDARY OUTCOMES:
HbA1c | at randomization, after 6, 12, and 18 months of treatment
insulin dose | at randomization, and after 3, 6, 12, and 18 months of treatment
adverse events | at randomization, and after 3, 6, 12, and 18 months of treatment
serum lipids | at randomization, and after 3, 6, 12, and 18 months of treatment
plasma CRP | at randomization, and after 3, 12, and 18 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Martin, MD, Principal Investigator — DDZ Deutsches Diabetes Zentrum, Düsseldorf, Germany
Locations (12):
- Germany (12):
  - Diabetes-Zentrum Mergentheim, Bad Mergentheim
  - Gemeinschaftskrankenhaus Havelhöhe, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Praxis Dr. Friedhelm Schmitten, Bestwig-Ramsbeck
  - St. Antonius Krankenhaus, Med. Klinik, Cologne
  - DDZ Deutsches Diabetes Zentrum, Düsseldorf
  - St. Josefs Krankenhaus, Heidelberg
  - Praxisklinik Leipzig, Leipzig
  - Praxis Dr. Gerhard Willms, Leverkusen
  - Praxis Dr. Heinz-Georg Ley, Marl
  - Diabetologische Schwerpunktpraxis, Angiologie, Münster
  - Praxis Dr. Werner Stürmer, Würzburg

REFERENCES:
- [Derived] Kolb H, Luckemeyer K, Heise T, Herder C, Schloot NC, Koenig W, Heinemann L, Martin S; DIATOR Study Group. The systemic immune network in recent onset type 1 diabetes: central role of interleukin-1 receptor antagonist (DIATOR Trial). PLoS One. 2013 Aug 26;8(8):e72440. doi: 10.1371/journal.pone.0072440. eCollection 2013. PMID 23991111
- [Derived] Strom A, Kolb H, Martin S, Herder C, Simon MC, Koenig W, Heise T, Heinemann L, Roden M, Schloot NC; DIATOR Study Group. Improved preservation of residual beta cell function by atorvastatin in patients with recent onset type 1 diabetes and high CRP levels (DIATOR trial). PLoS One. 2012;7(3):e33108. doi: 10.1371/journal.pone.0033108. Epub 2012 Mar 20. PMID 22448235
- [Derived] Martin S, Herder C, Schloot NC, Koenig W, Heise T, Heinemann L, Kolb H; DIATOR Study Group. Residual beta cell function in newly diagnosed type 1 diabetes after treatment with atorvastatin: the Randomized DIATOR Trial. PLoS One. 2011 Mar 11;6(3):e17554. doi: 10.1371/journal.pone.0017554. PMID 21412424